CLINICAL TRIAL: NCT02208895
Title: Correlation of In-lab Pleural Fluid Glucose Measurements With a Finger Stick Glucometer and Portable Point of Care Testing Device (i-STAT).
Brief Title: iSTAT Comparison Study, IRB3785
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 3785; VAMC OKC (Other: VAMC OKC)
Record Dates: First submitted 2014-07-31; First posted 2014-08-05 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Pleural Effusions
Keywords: pleural; glucose; glucometer; i-STAT
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Pleural fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- iSTAT Study Group: Measure glucose of pleural fluid via glucometer, in the laboratory, and using the iSTAT device to see if the three methods give a similar reading or not.

SUMMARY:
Pleural fluid glucose levels measured with bed-side point of care methods such as finger stick glucometers and I-STAT device correlate with the traditional in-lab testing methods.

DETAILED DESCRIPTION:
This is a prospective study which will identify patients in VAMC with a diagnosis of pleural effusion and undergoing diagnostic thoracentesis.The investigators plan to analyze the two bedside point-of-care fluid glucose testing methods (I- STAT device and finger stick glucometer) to measure pleural fluid glucose levels. The results obtained from these two methods will be compared to the traditionally in lab measured pleural fluid glucose levels.

ELIGIBILITY:
Inclusion Criteria:

* any patient 18 to 99 year old with a diagnosis of pleural effusion and undergoing a diagnostic thoracentesis.

Exclusion Criteria:

* Inability to provide informed consent by the patient or the surrogate to enroll for the planned study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pleural effusions
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-02; Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Correlation of pleural fluid glucose measured with a glucometer and the I-STAT with the pleural fluid glucose level measured in the Lab | <1 hour
  Primary outcome will be the inter-assay precision of the finger stick glucometer and the I-STAT device as compared to the Gold standard in lab testing of pleural glucose.This will be done using the Bland-Altman plot.

SECONDARY OUTCOMES:
Intra assay precision of pleural fluid glucose measured with a glucometer and with an I-STAT device. | < 1hour
  assessment of intra assay precision of of 2 measurements of pleural fluid glucose done by the glucometer as well as the ISTAT device .

CONTACTS AND LOCATIONS:
Overall Officials: Houssein Youness, MD, Principal Investigator — OUHSC
Locations (1):
- VAMC OKC, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data may only be shared upon review of OUHSC Legal office and IRB. Data sharing agreement required. Contact research@ouhsc.edu to initiate data requests. No personally identifiable data will be shared.